CLINICAL TRIAL: NCT01269177
Title: Mortality and Risk Factors in Patients With Acute Cardiogenic Pulmonary Edema: a Multicentric, Observational, Prospective Study
Acronym: ACPE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Milan (Other)
Responsible Party: Roberto Cosentini, MD, Fondazione IRCCS Ospedale Maggiore Policlinico, Mangiagalli, Regina Elena
Other Study IDs: ACPE.IT
Record Dates: First submitted 2011-01-03; First posted 2011-01-04 (Estimated); Last update posted 2011-01-04 (Estimated); Status verified 2010-10

CONDITIONS: Pulmonary Edema; Respiratory Insufficiency
Keywords: ACPE; Acute respiratory failure; Non invasive ventilation; acute cardiogenic pulmonary edema
MeSH Terms: conditions — Pulmonary Edema; Respiratory Insufficiency | interventions — Noninvasive Ventilation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Patients with acute cardiogenic pulmonary edema
  Interventions: Device: Non invasive ventilation

INTERVENTIONS:
Device: Non invasive ventilation — Indications for the use of NIV are at least one of the following:
  * Respiratory Rate ≥ 30 bpm
  * PaO2/FiO2 < 200
  * pH < 7.35 and PaCO2 > 45 mmH
  Contraindications for the use of NIV are at least one of the following:
  * Coma
  * Hemodynamic instability / shock
  * Lack of compliance
  Indications for endotracheal intubation (ETI) are at least one of the following:
  * Respiratory or cardiac arrest
  * Coma
  * Hemodynamic instability

SUMMARY:
The purpose of this study is to define the current treatment of patients ospitalized with acute cardiogenic pulmonary edema. Clinical and laboratory data collected in the Emergency Department will used to investigate the primary outcome (mortality) and risk factors related to the primary outcome.

DETAILED DESCRIPTION:
ACPE is a common cause of presentation to the Emergency Department (ED). Early recognition of high-risk patients could help in better locating human and technical resources and in deciding adequate treatment and site of care.

The investigators planned a real life, multicentric, prospective, web-based observational study performed in Italian Emergency Departments.

The investigators enroll consecutive patients admitted to the Emergency Department with acute cardiogenic pulmonary edema, that is defined as all the following: respiratory distress, bilateral rales and congestion on chest X-ray.

Demographic, clinical and laboratory findings are collected on admission and during hospitalization to evaluate mortality and risk factors related to mortality.

ELIGIBILITY:
Inclusion Criteria:

all of the following:

* age ≥ 18
* acute-onset dyspnea
* widespread pulmonary rales
* pulmonary congestion on chest X- ray plus one of the following:
* respiratory distress
* respiratory rate ≥ 30
* emogasanalysis: pH < 7.35 and pCO2 > 45 mmHg in Venturi-Mask 50%

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the Emergency Department with acute cardiogenic pulmonary edema
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2009-05

PRIMARY OUTCOMES:
mortality | Discharge from hospital

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Cosentini, MD, Study Chair — Ospedale Maggiore Policlinico Mangiagalli e Regina Elena
Locations (1):
- Fondazione IRCCS Ospedale Maggiore Policinico, Mangiagalli e Regina Elena, Milan, Italy, Italy

REFERENCES:
- [Background] Cosentini R, Aliberti S, Bignamini A, Piffer F, Brambilla AM. Mortality in acute cardiogenic pulmonary edema treated with continuous positive airway pressure. Intensive Care Med. 2009 Feb;35(2):299-305. doi: 10.1007/s00134-008-1281-7. Epub 2008 Sep 20. PMID 18807009
- See also: Related Info — http://www.acpe.it